CLINICAL TRIAL: NCT04177888
Title: Effect of Hot Pack on Labor Pain, Duration of Labor, and Satisfaction of Primigravidae Women in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Halimah Ali Alshahrani, Midwife, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: E-19-4027
Record Dates: First submitted 2019-11-22; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Labor Pain; Duration of Labor; Satisfaction
Keywords: Hot pack, Labor pain, Duration of labor, Satisfaction, Primigravid women
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: experimental group received who received hot pack, which was a single-use pack filled with magnesium sulfate and water, squeezed between the hands to activate the warming effect, applied to the lower back area. The control group received routine care including Entonox.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (Experimental): Experimental group with 45 participants, received hot pack, which was a single-use pack filled with magnesium sulfate and water, squeezed between the hands to activate the warming effect, applied to the lower back area for 30 minutes followed by 10 minutes rest then again applied for 30 minutes. This procedure was repeated till delivery.
  Interventions: Device: Hot Pack
- Control group (No Intervention): Control group with 46 participants received the hospital routine care that included Entonox inhalation as optional labor pain management.

INTERVENTIONS:
Device: Hot Pack — It is a single-use pack filled with magnesium sulfate and water, which was squeezed between the hands to activate their warming effect. The temperature ranges between 40°C to 50°C, which is safe to use. Thus, it provided a consistent heat therapy for up to 30 minutes. They can be used directly on the skin or covered with gauze to avoid direct skin contact. Applied to the lower back area for 30 minutes, followed by 10 minutes rest between each hot pack application, then it was reapplied for another 30 minutes. This procedure was repeated till delivery.
  Arms: Experimental group

SUMMARY:
The study aimed at determining the effect of hot pack on labor pain reduction and the duration of labor in comparison with routine care. Further, the study also aimed at determining the women's satisfaction with the use of hot pack and with routine care

with hypotheses: H1: Primigravid women who received hot pack in the active phase of labor will have a significantly lower mean labor pain score than those who received routine care.

H2: Primigravid women who received hot pack in the active phase of labor will have significantly shorter mean labor duration than those who received routine care.

DETAILED DESCRIPTION:
Childbirth pain is the severest type of pain that women experience in their life. Therefore, effective management of labor pain is essential. There are various methods to control childbirth pain: pharmacological and non-pharmacological such as Entonox and heat therapy respectively. In most Saudi Arabian hospitals, Entonox is used as routine care, while non- pharmacological agents are rarely used. Various forms of heat therapy are effective in labor pain reduction and shortening the duration of labor. There is a dearth for studies that compare the effectiveness of the hot pack with routine care that includes use of Entonox.

Objectives

* To determine the effect of the hot pack on labor pain reduction among primigravid women.
* To determine the effect of the hot pack on the duration of labor among primigravid women.
* To determine the satisfaction of primigravid women regarding hot pack and routine care.

Methods The study was conducted in Armed Forces Hospital Southern Region, with randomized sample of 91 primigravidae with normal pregnancy in active phase of first stage of labor, with cervical dilatation of 6 - 8 cm. This randomized controlled trial consisted of two groups: the experimental group (n = 45) who received hot pack. The control group (n = 46) received routine care including Entonox. Labor pain was assessed by Visual Analogue Scale for pain intensity (VAS); duration of labor was measured by the WHO modified partograph, and women's satisfaction was assessed using a satisfaction scale. Following eligibility assessment, participants were selected and allocated to the groups randomly. After obtaining the written informed consent, the initial assessment was done; the experimental group received hot pack, and the control group received routine care until delivery. The baseline pain score was assessed before the intervention and every 30 minutes after the intervention until delivery. The duration of labor was assessed using the WHO Partograph. The women reported satisfaction two hours post-delivery using the satisfaction scale.

Results:

Before the intervention, the experimental and control group did not differ statistically in terms of labor pain score (p = .820). Post-intervention, the labor pain score was significantly lower in the experimental groups (p ≤ 0.05) compared to the control group at 30, 60, 90, 120, 150 and 210 minutes. The duration of the first, second, and third stages of labor was not significantly different among both groups (p ≥ 0.05). The overall mean satisfaction scores were significantly higher in the experimental group compared to the control group (p ≤ 0.05), the mean scores of two items, one on happiness with the care received, and the other with the delivery experience were not significantly different between both groups (p ≥ 0.05).

Conclusion:

Heat therapy, such as the hot pack is a non-pharmacological method for labor pain management. Heat therapy is effective in reducing labor pain. Although it has been not effective in shortening the duration of labor, women are satisfied with the use of hot pack. This finding could be useful in formulating policies regarding implementation of the non-pharmacological methods for labor pain management. It is essential to educate healthcare professionals regarding the benefits of heat therapy even before implementing a change.

ELIGIBILITY:
Inclusion Criteria:

Saudi primigravid women who:

* Have normal term pregnancy (37 to 42 weeks) and have normal onset of labor.
* Are in the active phase of the first phase of labor with cervical dilatation of 6 cm and above and admitted to labor and delivery unit at Armed Forces Hospital Southern Region (AFHSR).
* Agreed to receive routine care including Entonox inhalation or to hot pack as pain management method during labor.

Exclusion Criteria:

Saudi primigravid women who:

* Are with contraindications for hot packs (fever, area injury or inflammation, skin infection, eczema, bleeding, Deep Vein Thrombosis (DVT), edema and poor thermal regulation),
* Have complicated pregnancy (polyhydramnios, oligohydramnios, decreased fetal movement, Intrauterine Growth Restriction (IUGR), Intrauterine Fetal Death (IUFD), Ante Partum Hemorrhage (APH), history of infertility, gestational hypertension, gestational diabetes, placenta previa, and placental abruption).
* Have medical conditions such as asthma, pneumonia, chest infection, chronic disease; such as cardiovascular disease, hypertension, and diabetes.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-25 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Partograph | 1-8 hours during labor
  The partograph is a universal tool to assess the progress of labor, it included graphical information with three main components; fetal condition, the progress of labor, and maternal condition. The researcher used the progress of labor component in the partograph to calculate the duration of labor in minutes.
Satisfaction Scale | Used two hours post delivery for both group to assess women's satisfaction regarding the intervention and routine care
  A Likert-type scale with five points. The scale descriptions: (5) very satisfied, (4) satisfied, (3) neither satisfied nor dissatisfied, (2) dissatisfied, and (1) very dissatisfied
Visual Analogue Scale for Pain Intensity (VAS) "change" is being assessed | 1-8 hours during labor
  It is a one item scale that involves a horizontal or vertical line which starts either with 0 to 10 cm. Zero is no pain and 10 is the worst or intolerable pain. the interpretation is zero no pain, 1 - 3 cm mild pain, 4 - 6 cm moderate pain, 7 - 9 cm severe pain, and 10 cm intolerable or worst pain possible.
  baseline labor pain assessed, then VAS used every 30 minutes to assess labor pain till delivery

CONTACTS AND LOCATIONS:
Overall Officials: Halimah A Alshahrani, Master, Principal Investigator — KSU, AFHSR
Locations (1):
- KSU, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
individual participant data (IPD) will not be shared